CLINICAL TRIAL: NCT05945043
Title: Continuation Of a Study to Investigate the Effect of Thoracocentesis on Neural Respiratory Drive in Pleural Effusion (COSINE)
Brief Title: Continuation Of a Study to Investigate the Effect of Thoracocentesis on Neural Respiratory Drive in Pleural Effusion
Acronym: COSINE
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322762
Record Dates: First submitted 2023-06-07; First posted 2023-07-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pleural Effusion
Keywords: Pleural effusion; Breathlessness; Neural respiratory drive; Neurophysiology
MeSH Terms: conditions — Pleural Effusion; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic pleural effuion: Patients with symptomatic unilateral pleural effusion of any cause who will be undergoing pleural fluid removal via thoracocentesis, chest drain insertion or IPC drainage for relief of their breathlessness.
  Interventions: Other: Surface parasternal eletromyogram; Other: Surface diaphragm electromyogram; Other: Parasternal muscle ultrasound; Other: Breathlessness assessment

INTERVENTIONS:
Other: Surface parasternal eletromyogram — The surface parasternal EMG of participants will be measured pre, immediately post and at days 1 and 7 following pleural fluid removal
Other: Surface diaphragm electromyogram — The ipsilateral and contralateral surface diaphragm EMG of participants will be measured pre and immediately post pleural fluid removal
Other: Parasternal muscle ultrasound — The thickness of the parasternal intercostal muscle of participants will be measured using thoracic ultrasound pre and immediately post pleural fluid removal
Other: Breathlessness assessment — The VAS breathlessness score and Dyspnoea-12 questionnaire of participants will be measured pre, immediately post and at days 1 and 7 following pleural fluid removal

SUMMARY:
The aim of this study is to better understand the relationship between pleural effusions and breathlessness in patients with unilateral pleural effusions and breathlessness who require pleural fluid removal for its management.

DETAILED DESCRIPTION:
This study will involve 124 adult patients who are breathlessness with pleural effusions. They will be recruited from a single UK centre over an 18-month period.

After being informed about the study, all patients giving written informed consent will undergo a baseline assessment when they first come to have their fluid drained. The investigators will record information about them and their disease. The investigators will take measurements of their breathlessness, their breathing muscles, and the electrical activity from the brain to those muscles. These will be taken at the start and end of drainage, as well as 1 day and 7 days after. The investigators will use this information to look for links between the effect of pleural effusions and its removal on the electrical activities of the breathing muscles and patients' breathlessness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Has a unilateral pleural effusion AND

  1. require thoracocentesis OR
  2. chest drain insertion (main study only) OR
  3. has an IPC in situ (main study only)

Exclusion Criteria:

* Inability to consent
* Any contraindications to the proposed pleural procedure
* Haemodynamic or clinical instability that precludes from the safe completion of required pre-procedural measurements
* Inability to identify surface landmarks for surface EMG electrode placement
* Past medical history of diaphragmatic paralysis (diaphragm sub study only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with unilateral pleural effusions requiring pleural fluid removal via thoracocentesis, chest drain insertion or IPC drainage for management of their breathlessness.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Neural respiratory drive (as measured by surface parasternal EMG) at 24 hours post pleural fluid removal | 24 hours
  Neural respiratory drive index (as measured by surface parasternal EMG)
Patient reported breathlessness (as measured by VAS dyspnoea score) at 24 hours post pleural fluid removal | 24 hours
  VAS dyspnoea score

SECONDARY OUTCOMES:
Neural respiratory drive (as measured by surface parasternal EMG) at other time points post pleural fluid removal | pre procedure, immediately post procedure and daily up to 7 days
  Neural respiratory drive index (as measured by surface parasternal EMG)
Patient reported breathlessness (as measured by VAS dyspnoea score) at other time points post pleural fluid removal | pre procedure, immediately post procedure and daily up to and 7 days
  VAS dyspnoea score
The effect on exercise capacity of pleural fluid removal. | pre procedure, immediately post procedure, 1 day and 7 days
  6 min walk test
Pleural effusion characteristics as measured by thoracic ultrasound | immediately post procedure, 1 day and 7 days
  Thoracic ultrasound
To determine the acceptability of incorporating surface parasternal EMG measurement as part of routine clinical practice to patients and clinicians | peri-procedural
  Qualitative feedback form
Neural respiratory drive (as measured by surface diaphragm EMG) of the ipsilateral hemidiaphragm following thoracocentesis | peri-procedural
  Neural respiratory drive index (as measured by surface diaphragm EMG)
Ipsilateral hemidiaphragm morphology and movement as measured by thoracic ultrasound. | peri-procedural
  Thoracic ultrasound
Neural respiratory drive (as measured by surface diaphragm EMG) of the contralateral hemidiaphragm following thoracocentesis | peri-procedural
  Neural respiratory drive index (as measured by surface diaphragm EMG)
Contralateral hemidiaphragm morphology and movement as measured by thoracic ultrasound. | peri-procedural
  Thoracic ultrasound
Parasternal intercostal muscle thickness as measured by thoracic ultrasound following pleural fluid removal | peri-procedural
  Thoracic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Murphy, MBBS BSc, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhatnagar R, Maskell N. The modern diagnosis and management of pleural effusions. BMJ. 2015 Sep 8;351:h4520. doi: 10.1136/bmj.h4520. No abstract available. PMID 26350935
- [Result] Marel M, Zrustova M, Stasny B, Light RW. The incidence of pleural effusion in a well-defined region. Epidemiologic study in central Bohemia. Chest. 1993 Nov;104(5):1486-9. doi: 10.1378/chest.104.5.1486. PMID 8222812
- [Result] Thomas R, Jenkins S, Eastwood PR, Lee YC, Singh B. Physiology of breathlessness associated with pleural effusions. Curr Opin Pulm Med. 2015 Jul;21(4):338-45. doi: 10.1097/MCP.0000000000000174. PMID 25978627
- [Result] Estenne M, Yernault JC, De Troyer A. Mechanism of relief of dyspnea after thoracocentesis in patients with large pleural effusions. Am J Med. 1983 May;74(5):813-9. doi: 10.1016/0002-9343(83)91072-0. PMID 6837605
- [Result] Psallidas I, Yousuf A, Talwar A, Hallifax RJ, Mishra EK, Corcoran JP, Ali N, Rahman NM. Assessment of patient-reported outcome measures in pleural interventions. BMJ Open Respir Res. 2017 Jul 3;4(1):e000171. doi: 10.1136/bmjresp-2016-000171. eCollection 2017. PMID 28883922
- [Result] Muruganandan S, Azzopardi M, Thomas R, Fitzgerald DB, Kuok YJ, Cheah HM, Read CA, Budgeon CA, Eastwood PR, Jenkins S, Singh B, Murray K, Lee YCG. The Pleural Effusion And Symptom Evaluation (PLEASE) study of breathlessness in patients with a symptomatic pleural effusion. Eur Respir J. 2020 May 14;55(5):1900980. doi: 10.1183/13993003.00980-2019. Print 2020 May. PMID 32079642
- [Result] Nishino T. Dyspnoea: underlying mechanisms and treatment. Br J Anaesth. 2011 Apr;106(4):463-74. doi: 10.1093/bja/aer040. Epub 2011 Mar 4. PMID 21378105
- [Result] Light RW, Stansbury DW, Brown SE. The relationship between pleural pressures and changes in pulmonary function after therapeutic thoracentesis. Am Rev Respir Dis. 1986 Apr;133(4):658-61. doi: 10.1164/arrd.1986.133.4.658. PMID 3963629
- [Result] Skaarup SH, Lonni S, Quadri F, Valsecchi A, Ceruti P, Marchetti G. Ultrasound Evaluation of Hemidiaphragm Function Following Thoracentesis: A Study on Mechanisms of Dyspnea Related to Pleural Effusion. J Bronchology Interv Pulmonol. 2020 Jul;27(3):172-178. doi: 10.1097/LBR.0000000000000627. PMID 31651544
- [Result] Fitzgerald DB, Muruganandan S, Peddle-McIntyre CJ, Lee YCG, Singh B. Ipsilateral and contralateral hemidiaphragm dynamics in symptomatic pleural effusion: The 2nd PLeural Effusion And Symptom Evaluation (PLEASE-2) Study. Respirology. 2022 Oct;27(10):882-889. doi: 10.1111/resp.14307. Epub 2022 Jun 7. PMID 35672271
- [Result] De Troyer A, Kirkwood PA, Wilson TA. Respiratory action of the intercostal muscles. Physiol Rev. 2005 Apr;85(2):717-56. doi: 10.1152/physrev.00007.2004. PMID 15788709
- [Result] Decramer M. Hyperinflation and respiratory muscle interaction. Eur Respir J. 1997 Apr;10(4):934-41. PMID 9150337
- [Result] Jolley CJ, Moxham J. A physiological model of patient-reported breathlessness during daily activities in COPD. Eur Respir Rev. 2009 Jun;18(112):66-79. doi: 10.1183/09059180.00000809. PMID 20956127
- [Result] Finucane KE, Panizza JA, Singh B. Efficiency of the normal human diaphragm with hyperinflation. J Appl Physiol (1985). 2005 Oct;99(4):1402-11. doi: 10.1152/japplphysiol.01165.2004. Epub 2005 Jun 16. PMID 15961606
- [Result] De Troyer A, Wilson TA. Effect of acute inflation on the mechanics of the inspiratory muscles. J Appl Physiol (1985). 2009 Jul;107(1):315-23. doi: 10.1152/japplphysiol.91472.2008. Epub 2009 Mar 5. PMID 19265064
- [Result] Wallbridge P, Hew M, Parry SM, Irving L, Steinfort D. Reduction of COPD Hyperinflation by Endobronchial Valves Improves Intercostal Muscle Morphology on Ultrasound. Int J Chron Obstruct Pulmon Dis. 2020 Dec 7;15:3251-3259. doi: 10.2147/COPD.S282829. eCollection 2020. PMID 33324048
- [Result] Lalley PM. Respiration - Neural Control. In: Binder MD, Hirokawa N, Windhorst U, editors. Encyclopedia of Neuroscience. Berlin, Heidelberg: Springer Berlin Heidelberg; 2009. p. 3433-41.
- [Result] Killian KJ, Gandevia SC, Summers E, Campbell EJ. Effect of increased lung volume on perception of breathlessness, effort, and tension. J Appl Physiol Respir Environ Exerc Physiol. 1984 Sep;57(3):686-91. doi: 10.1152/jappl.1984.57.3.686. PMID 6490457
- [Result] Adams L, Lane R, Shea SA, Cockcroft A, Guz A. Breathlessness during different forms of ventilatory stimulation: a study of mechanisms in normal subjects and respiratory patients. Clin Sci (Lond). 1985 Dec;69(6):663-72. doi: 10.1042/cs0690663. PMID 3933895
- [Result] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Result] Jolley CJ, Luo YM, Steier J, Reilly C, Seymour J, Lunt A, Ward K, Rafferty GF, Polkey MI, Moxham J. Neural respiratory drive in healthy subjects and in COPD. Eur Respir J. 2009 Feb;33(2):289-97. doi: 10.1183/09031936.00093408. Epub 2008 Oct 1. PMID 18829678
- [Result] Reilly CC, Ward K, Jolley CJ, Lunt AC, Steier J, Elston C, Polkey MI, Rafferty GF, Moxham J. Neural respiratory drive, pulmonary mechanics and breathlessness in patients with cystic fibrosis. Thorax. 2011 Mar;66(3):240-6. doi: 10.1136/thx.2010.142646. Epub 2011 Feb 1. PMID 21285244
- [Result] Jolley CJ, Luo YM, Steier J, Rafferty GF, Polkey MI, Moxham J. Neural respiratory drive and breathlessness in COPD. Eur Respir J. 2015 Feb;45(2):355-64. doi: 10.1183/09031936.00063014. Epub 2014 Oct 16. PMID 25323229
- [Result] Reilly CC, Jolley CJ, Ward K, MacBean V, Moxham J, Rafferty GF. Neural respiratory drive measured during inspiratory threshold loading and acute hypercapnia in healthy individuals. Exp Physiol. 2013 Jul;98(7):1190-8. doi: 10.1113/expphysiol.2012.071415. Epub 2013 Mar 15. PMID 23504646
- [Result] MacBean V, Hughes C, Nicol G, Reilly CC, Rafferty GF. Measurement of neural respiratory drive via parasternal intercostal electromyography in healthy adult subjects. Physiol Meas. 2016 Nov;37(11):2050-2063. doi: 10.1088/0967-3334/37/11/2050. Epub 2016 Oct 25. PMID 27779132
- [Result] Murphy PB, Kumar A, Reilly C, Jolley C, Walterspacher S, Fedele F, Hopkinson NS, Man WD, Polkey MI, Moxham J, Hart N. Neural respiratory drive as a physiological biomarker to monitor change during acute exacerbations of COPD. Thorax. 2011 Jul;66(7):602-8. doi: 10.1136/thx.2010.151332. Epub 2011 May 19. PMID 21597112
- [Result] Reilly CC, Jolley CJ, Elston C, Moxham J, Rafferty GF. Measurement of parasternal intercostal electromyogram during an infective exacerbation in patients with cystic fibrosis. Eur Respir J. 2012 Oct;40(4):977-81. doi: 10.1183/09031936.00163111. Epub 2012 Jan 20. PMID 22267769
- [Result] Lin L, Guan L, Wu W, Chen R. Correlation of surface respiratory electromyography with esophageal diaphragm electromyography. Respir Physiol Neurobiol. 2019 Jan;259:45-52. doi: 10.1016/j.resp.2018.07.004. Epub 2018 Jul 21. PMID 30041019
- [Result] Bellani G, Bronco A, Arrigoni Marocco S, Pozzi M, Sala V, Eronia N, Villa G, Foti G, Tagliabue G, Eger M, Pesenti A. Measurement of Diaphragmatic Electrical Activity by Surface Electromyography in Intubated Subjects and Its Relationship With Inspiratory Effort. Respir Care. 2018 Nov;63(11):1341-1349. doi: 10.4187/respcare.06176. PMID 30389829
- [Result] Luiso D, Villanueva JA, Belarte-Tornero LC, Fort A, Blazquez-Bermejo Z, Ruiz S, Farre R, Rigau J, Marti-Almor J, Farre N. Surface respiratory electromyography and dyspnea in acute heart failure patients. PLoS One. 2020 Apr 29;15(4):e0232225. doi: 10.1371/journal.pone.0232225. eCollection 2020. PMID 32348374
- [Result] Korczynski P, Gorska K, Konopka D, Al-Haj D, Filipiak KJ, Krenke R. Significance of congestive heart failure as a cause of pleural effusion: Pilot data from a large multidisciplinary teaching hospital. Cardiol J. 2020;27(3):254-261. doi: 10.5603/CJ.a2018.0137. Epub 2018 Nov 8. PMID 30406935
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180